CLINICAL TRIAL: NCT01171560
Title: Prospective Randomized Clinical Trial for Single-Lung-Ventilation Comparing Double-Lume Tube and the EZ-Blocker®
Brief Title: Evaluation of the EZ Blocker
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Department of Cardio-, Thoracic- and Vascular- Anesthesia, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 096/2010
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-05

CONDITIONS: Intubation; Thoracic Surgery; One-lung Ventilation
Keywords: EZ Blocker; Double-lumen Tube; Airway; thoracic surgery; time for intubation; blind insertion; conditions of surgery; postoperative sore throat; postoperative hoarseness
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EZ Blocker (Active Comparator): Patients assigned to the EZ group will be intubated using a conventional tube in an adequate size as it is standard of care and single lung ventilation will be provided using the EZ-Blocker.
  Interventions: Procedure: endotracheal intubation
- Double lumen tube (Active Comparator): The patients assigned to the "double lume tube" group will be intubated using the double lume tube in an adequate size as it is standard of care.
  Interventions: Procedure: endotracheal intubation

INTERVENTIONS:
Procedure: endotracheal intubation — The patients will be randomized to one of two groups: EZ Blocker or conventional double lume tube. After induction of anesthesia, intubation using respective device will be performed in dorsal position.

SUMMARY:
In anesthetized patients the airway needs to be secured due to lack of protective reflexes. Golden standard is the endotracheal intubation. In patients undergoing lung surgery single lung ventilation is essential. In these cases a double lume tube is commonly used. The double lume tube has a proximal tracheal and a distal bronchial end reaching into the left or the right side of the lung dependant of the model of the tube. Thus it is possible to operate on one collapsed side of the lung while ventilating the other side.

Due to length and stiffness resulting of the construction of the device more side effects than after intubation with a conventional single lumen tube is expected. Possible side effects may be bleeding, swelling, sore throat or croakiness.

The EZ-Blocker is a new device promising to overcome these side effects. The EZ-Blocker is a device placing a balloon into one bronchus to be able to provide single lung ventilation like the double lume tube. However, the EZ-Blocker is a catheter pushed through a conventional single lume tube after intubation with a hook on one and a balloon on the other distal end. The hook prevents the device from being pushed too far to be able to harm the lung. Inside the EZ-Blocker is a small lumen able to deflate the lung which is blocked with the balloon. The device is easily positioned using a bronchoscope and when the anaesthesiologists confirmed the correct position of the device, the balloon can be inflated and deflated as needed.

Due to the easier approach the investigators expect less side effects as mentioned earlier using the EZ-Blocker compared to the double lume tube. As well the stress caused by intubation may be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* thoracic surgery with requiring single lung ventilation in lateral position
* ASA Status 1-3
* Oral and written consent to participation
* Age 18- 90

Exclusion Criteria:

* Contraindications against placing a double lume tube, like tracheal lesions, etc.
* Thoracic surgery within the last four weeks
* Any form of infection (Pneumonia, Pleural empyema) or suspected Tbc
* BMI higher than 45
* Patients with a previous diagnoses or suspected difficult airway

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-07 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Time from intubation to ventilation: | 5 minutes
  is intubation and achieving lung separation faster using a conventional double-lung-tube or using the EZ-Blocker ?

SECONDARY OUTCOMES:
postoperative sore throat or croakiness | 2 minutes
  Documentation of sore throat and croakiness by questioning the patients the day after surgery
resistance to dislocation | 10 minutes
  Which device, double-lung-tube or EZ-Blocker, is more resistant to dislocation in endotracheal/endobronchial position, especially when the patient is moved from dorsal to lateral position?
Peripheral oxygen saturation (SpO2) | 3 hours
  Decrease of Peripheral oxygen saturation (SpO2) (in min) under 90% during the hole surgery

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Ruetzler K, Grubhofer G, Schmid W, Papp D, Nabecker S, Hutschala D, Lang G, Hager H. Randomized clinical trial comparing double-lumen tube and EZ-Blocker for single-lung ventilation. Br J Anaesth. 2011 Jun;106(6):896-902. doi: 10.1093/bja/aer086. Epub 2011 Apr 14. PMID 21493621